CLINICAL TRIAL: NCT05193123
Title: Psychological Trauma and Resilience After ICU Stay in Patients Treated With Mechanical Ventilation for Severe Critical Illness: the Multicenter, Prospective, Observational RESIREA Study
Brief Title: Psychological Trauma and Resilience After Critical Illness
Acronym: RESIREA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MR_Resirea
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Acute Respiratory Failure; Shock
Keywords: critical illness; mechanical ventilation; shock; post-traumatic stress disorder; resilience; psychological trauma
MeSH Terms: conditions — Shock; Critical Illness; Stress Disorders, Post-Traumatic; Psychological Trauma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Critically ill patients experience a severe physical disease, associated with a psychotrauma, which may lead to post-traumatic stress disorder (17 to 30% of patients after critical illness) and persistent symptoms of anxiety and depression. RESIREA study will study psychodrama, resilience and factors associated with resilience in patients previously included in the NUTRIREA-3 randomized controlled trial designed to compare standard calorie and protein feeding complying with guidelines to low-calorie low-protein feeding in a well-defined group of severely ill ICU patients requiring at least MV and vasoactive drugs.

DETAILED DESCRIPTION:
Social demographic data (gender, age, marital status, psychological information and medical background) and medical data (severity of the disease, duration of ICU stay, SOFA score) will be collected, as for the NUTRIREA-3 trial.

Before leaving the ICU, patient who agreed to participate to the NUTRIREA 3 study were asked to participate to the RESIREA study.

Patients will be called by phone by a psychologist 3 months after their inclusion in the NUTRIREA-3 trial to complete the SF-36 score. Then, they will be asked to confirm their participation to the RESIREA study by completing four additional questionnaires (post-trauma stress disorder: IES-R; Resilience: CD-RISC; Social support: MSPSS; Perception of the disease: B-IPQ). If the patient does not respond to the phone call at the first time, he/she will be contacted again within a period of 2 weeks maximum (1 call/day). If the patient remains unreachable, he/she will be considered as lost for the study. Patients will be called again 12 months after their inclusion in the NUTRIREA-3 trial and will be asked to complete the five questionnaires (SF-36, IES-R, CD-RISC, MSPSS and B-IPQ).

During this last phone call, 40 patients will be asked to a third interview by phone. These patients will be spotted thanks to their score at the IES-R and CD-RISC. This interview of 30 to 45 minutes will be planned within 15 days after the T12 call and recorded. This semi structured interview will be lead by an experienced clinical psychologist and follow 4 main topics :

1. Experience of ICU's
2. Perception of the disease or/and post intensive care disorders
3. Difficulties and capacities of coping
4. Difficult events in the patient's life

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation started within the past 24 h, or started before ICU admission with ICU admission within the past 24 h, for an expected duration of at least 48 hours after inclusion
* Treatment with vasoactive agent for shock (adrenaline, dobutamine, or noradrenaline)
* Nutritional support expected to be started within 24 h after intubation
* Age older than 18 years
* Informed consent to participation in the study

Exclusion Criteria:

* Invasive mechanical ventilation started more than 24 hours earlier
* Specific nutritional needs, such as pre-existing long-term home enteral or parenteral nutrition, or for chronic bowel disease
* Dying patient, not-to-be-resuscitated order, or other treatment limitation decision at ICU admission
* Pregnancy, recent delivery, or lactation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients included in the NUTRIREA3 study will be contacted by phone calls to complete the quality of life scale (SF-36) 3 and 12 months after inclusion in the trial. Patients included in 24 of the 61 ICUs participating to the NUTRIREA-3 trial will be asked to participate to the RESIREA study at the 3-month phone call, by completing 4 additional questionnaires (IES-R, CD-RISC, MSPSS, B-IPQ), 3 and 12 month after their inclusion in the NUTRIREA-3 trial.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with post-traumatic disorders | 3 months after ICU stay
  IES-R scale

SECONDARY OUTCOMES:
Proportion of resilient patients | 3 and 12 months after ICU stay
  CD-RISC score > 80
proportion of patients with impaired Quality of life | 3 and 12 months after ICU stay
  SF-36 score
Proportion of patients with post-traumatic disorders | 12 months after ICU stay
  IES-R
Social support | 3 and 12 months after ICU stay
  IES-R
perception of the disease | 3 and 12 months after ICU stay
  MSPSS score

CONTACTS AND LOCATIONS:
Overall Officials: Jean REIGNIER, PhD, Principal Investigator — Nantes University Hospital
Locations (23):
- France (23):
  - CHU Amiens Picardie nord, Amiens
  - CHU Amiens Picardie sud, Amiens
  - CHU Angers, Angers
  - CH Angoulême, Angoulême
  - CH Annecy Genevois, Annecy
  - CH Argenteuil, Argenteuil
  - CHU Jean Minjoz, Besançon
  - CH de Béthune, Béthune
  - CH Chartres Louis Pasteur, Chartres
  - CHU Gabriel Montpided, Clermont-Ferrand
  - CH Dieppe, Dieppe
  - APHP - Hôpital Raymond Poincaré, Garches
  - CHD Vendée, La Roche-sur-Yon
  - CH du Mans, Le Mans
  - CH de Lens, Lens
  - CHR- Roger Salengro, Lille
  - Hôpital Edouard Herriot, Lyon
  - CHU de Nantes, Nantes
  - APHP - Hôpital Cochin, Paris
  - CH de Bigorre, Tarbes
  - CHRU Bretonneau, Tours
  - CHU de Valenciennes, Valenciennes
  - CHBA - Vannes Auray, Vannes